CLINICAL TRIAL: NCT02844881
Title: Phase I/IIa, Single-Arm, Open Study of Apatinib and MASCT in Patients With Advanced Solid Tumors
Brief Title: Study of Apatinib and MASCT in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First People's Hospital of Lianyungang (Other)
Collaborators: Hengrui Yuanzheng Bio-Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM-001
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Solid Tumors; Excluding T Cell Lymphoma
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apatinib+MASCT (Experimental): Apatinib+Multiple Antigens Specific Cellular Therapy(MASCT) in patients with advanced solid tumors,excluding T cell lymphoma
  Interventions: Drug: Apatinib; Biological: MASCT

INTERVENTIONS:
Drug: Apatinib — Apatinib 850 mg p.o. qd every 28 days until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Other Names: YN968D1
Biological: MASCT — Dendritic cells(DC) loaded with 17 antigens ih day 8, cytotoxic T lymphocytes ( CTL) induced by DC IV day 21-28, every 28 days until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends
  Other Names: Multiple Antigens Specific Cellular Therapy

SUMMARY:
The study is aimed to evaluate the efficacy and safety of Apatinib and MASCT in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Angiogenesis is a hallmark of cancer, together with vascular endothelial growth factor (VEGF) as one of the most important angiogenic drivers. Inhibitors targeting the VEGF/VEGFR-pathway have shown beneficial effects in many cancer patients, but they are transient and followed by fast regrowth. Similarly, the effectiveness of tumor immunotherapies has been limited by tumor-mediated escape mechanisms and immune suppression. By combining the two strategies, antiangiogenic immunotherapy offers the possibility to more vigorously inhibit tumor angiogenesis and promote an enduring immune-stimulatory milieu that leads to prolonged survival benefits in cancer patients.

Apatinib is a small-molecule tyrosine kinase inhibitor (TKI) that highly selectively binds to and strongly inhibits vascular endothelial growth factor receptor 2 (VEGFR-2). Apatinib has been demonstrated as monotherapy prolongs OS in patients with gastric or gastroesophageal junction adenocarcinoma after two or more lines of chemotherapy with moderate, reversible, and easily managed adverse events.

Multiple antigens specific cellular therapy (MASCT) is a new immunotherapy that dendritic cells(DC) was induced from autologous peripheral blood. The DC can then be loaded with 17 antigens and re-infused. In vitro, antigen-pulsed DC can stimulate autologous T-cell proliferation and induction of autologous specific cytotoxic T-cells(CTL)，similarly re-infused. The previous research data showed that MASCT had the modest overall response and less adverse effects for Hepatocellular Carcinoma patients.

The study is aimed to evaluate the efficacy and safety of Apatinib and MASCT in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically-confirmed, advanced (unresectable) solid tumors who have progressed on standard therapy.
2. With written informed consent signed voluntarily by patients themselves.
3. The time of between Patients enrollment and the end of other anti-tumors therapies≤1 month
4. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) of ≤ 2
5. At least one measurable lesion as defined by RECIST criteria 1.1 for solid tumors.
6. Life expectancy ≥6 months.
7. With normal cardiopulmonary function.
8. Patients have adequate organ function as defined by the following criteria:

   * Hemoglobin (HGB) ≥85g/L
   * Absolute neutrophil count (ANC) ≥1.0×109/L
   * White blood cell (WBC) ≥3.0×109/L
   * Platelet count ≥50×109/L
   * Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) of ≤2.5 upper normal limitation (UNL) or ≤5 UNL in case of liver metastasis
   * Alkaline phosphatase (ALP)≤2.5 UNL
   * Total bilirubin (TBil) of ≤1.5 UNL
   * Blood urea nitrogen (BUN) and Creatinine (Cr) of≤1.5 UNL
   * Albumin (ALB) ≥30g/L

Exclusion Criteria:

1. Pregnant or expecting to pregnant
2. Participated in other clinical trials before screening except of observational study.
3. Known allergic history of sodium citrate drugs.
4. Known history of organ transplant, including autologous bone marrow transplantation and peripheral stem cell transplantation.
5. Known active brain metastases as determined by CT or MRI evaluation.
6. The use of immunosuppressive drugs with current or 14 days before enrollment.
7. Know the period of systemic and continuous use of immunomodulatory agents (such as interferon, thymosin, traditional Chinese medicine) within 6 months.
8. Prior therapy with anti-programmed death-1 (anti-PD-1), anti-programmed cell death ligand 1 (anti-PD-L1), or anti-Cytotoxic T lymphocyte-associated antigen 4 (anti-CTLA-4) antibody (including any other antibody or drug specifically targeting T-cell co-stimulation).
9. Known history of primary immunodeficiency diseases.
10. Known history of tuberculosis.
11. Known active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
12. Patients with serious infection, hepatopathy, nephropathy, respiratory disease, cardiovascular disease or incontrollable diabetes, etc.
13. Patients have other malignant tumors within 5 years,excluding melanoma and carcinoma in situ of cervix.
14. Treatment with any anti-tumors agent within 28days of first administration of study treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | up to 2 years
  The incidence of treatment-related adverse events were graded with the use of the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival)
Overall Survival (OS) | From enrollment to death of patients. Estimated about 1 year.
  The length of time from enrollment until the time of death (OS, overall survival)
Objective Response Rate (ORR) | up to 2 years
  clinical response of treatment according to RESIST v1.1 criteria (ORR, objective response rate)
Disease Control Rate (DCR) | up to 2 years
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) based on RESIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- The First's People Hospital of Lianyungang, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided